CLINICAL TRIAL: NCT01269268
Title: Characterization and Evaluation of Diagnostic Biomarkers for Tuberculosis
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0213
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Active Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood and serum will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- active tuberculosis: active TB patients : diagnosed with TB through microbiologic examination
- healthy control: healthy control : no evidence of respiratory disease, no respiratory symptoms, and no history of close contact of active pulmonary TB patients

SUMMARY:
There was no sensitive and specific biomarker for tuberculosis infection, disease progression and predicting the prognosis of treatment. Therefore, the investigators aimed to investigate and evaluate the newer biomarker for the diagnosis of TB infection. To investigate the new biomarker for TB infection, the investigators will recruit the participants including active TB patients, healthy household contacts, healthy community control.

ELIGIBILITY:
Inclusion Criteria:

* active TB patients : diagnosed with active TB through the microbiologic examination, imaging findings
* healthy control : no history of TB treatment, no respiratory symptoms, no evidence of active infectious disease including TB on chest X-ray, no history of close contacts of active pulmonary TB patients

Exclusion Criteria:

* pregnant woman
* positive result of human immunodeficiency virus examination

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: active TB patients group : from the referred center TB care clinic healthy control : from the community sample
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05-14 (Actual); Study Completion 2014-05-14 (Actual)

PRIMARY OUTCOMES:
Characterization of antigens of Mycobacterium tuberculosis K strain for serodiagnosis of tuberculosis | 6months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea